CLINICAL TRIAL: NCT05233436
Title: A PHASE 1, OPEN-LABEL, DOSE ESCALATION AND EXPANSION STUDY OF PF-07265028 AS A SINGLE AGENT AND IN COMBINATION WITH SASANLIMAB EVALUATING THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND ANTI-TUMOR ACTIVITY OF PF-07265028 IN PARTICIPANTS WITH ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: PF-07265028 As Single Agent And In Combination With Sasanlimab in Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated based on internal business considerations and was not based on safety reasons
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4731001
Record Dates: First submitted 2022-01-06; First posted 2022-02-10 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors; Gastric Cancer; Gastroesophageal Junction Cancer; Urothelial Cancer; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinomas
Keywords: immunotherapy; advanced solid tumor; metastatic solid tumor; first in human; Gastric cancer; Gastroesophageal junction cancer; Urothelial Cancer; Non small cell lung cancer; Head and neck squamous cell carcinomas; SCCHN; NSCLC; Lung cancer; Hematopoietic progenitor kinase 1 inhibitor; HPK1 inhibitor
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1A Dose Escalation Monotherapy (Experimental): Participants will receive PF-07265028 at escalating dose levels.
  Interventions: Drug: PF-07265028
- Part 1B Dose Escalation Combination (Experimental): Participants will receive PF-07265028 at escalating dose levels in combination with sasanlimab fixed dose
  Interventions: Drug: PF-07265028; Biological: Sasanlimab
- Part 2A Dose Expansion Combination (SCCHN) (Experimental): Participants with squamous cell carcinoma of the head and neck (SCCHN) will receive PF-07265028 in combination with sasanlimab at the recommended dose from Part 1B
  Interventions: Drug: PF-07265028; Biological: Sasanlimab
- Part 2A Dose Expansion Combination (UC) (Experimental): Participants with urothelial cancer (UC) will receive PF-07265028 in combination with sasanlimab at the recommended dose from Part 1B
  Interventions: Drug: PF-07265028; Biological: Sasanlimab
- Part 2A Dose Expansion Combination (Gastric/GEJ) (Experimental): Participants with gastric/gastroesophageal junction cancer (Gastric/GEJ) will receive PF-07265028 in combination with sasanlimab at the recommended dose from Part 1B
  Interventions: Drug: PF-07265028; Biological: Sasanlimab
- Part 2A Dose Expansion Combination (NSCLC) (Experimental): Participants with non small cell lung cancer (NSCLC) will receive PF-07265028 in combination with sasanlimab at the recommended dose from Part 1B
  Interventions: Drug: PF-07265028; Biological: Sasanlimab
- Part 2A Dose Expansion Combination (selected tumor types) (Experimental): Participants with selected tumor types will receive PF-07265028 in combination with sasanlimab at the recommended dose from Part 1B
  Interventions: Drug: PF-07265028; Biological: Sasanlimab
- Part 2B Dose Expansion Monotherapy (selected tumor types) (Experimental): Participants with selected tumor types will receive PF-07265028 single agent at the recommended dose from Part 1A.
  Interventions: Drug: PF-07265028

INTERVENTIONS:
Drug: PF-07265028 — PF-07265028 will be administered orally
Biological: Sasanlimab — Administered subcutaneously
  Other Names: PF-06801591
  Arms: Part 1B Dose Escalation Combination; Part 2A Dose Expansion Combination (Gastric/GEJ); Part 2A Dose Expansion Combination (NSCLC); Part 2A Dose Expansion Combination (SCCHN); Part 2A Dose Expansion Combination (UC); Part 2A Dose Expansion Combination (selected tumor types)

SUMMARY:
The purpose of this study is to assess the safety and effects of PF-07265028 as monotherapy and in combination with sasanlimab.

The study aims to identify the maximum tolerated dose (MTD) of PF-07265028 as monotherapy; evaluate the clinical activity of monotherapy and combination; and select the recommended dose of PF-07265028 monotherapy and in combination for potential further studies and development.

The study contains 2 parts, Dose Escalation (Part 1) to determine the recommended dose of PF-07265028 as single agent and in combination, followed by Dose Expansion (Part 2) in selected tumor types at the recommended dose.

It is expected that most participants will take part in this study for up to 1 year with six on-site visits in the first month and then at least twice every subsequent month while they are on treatment.

DETAILED DESCRIPTION:
The purpose of this first-in-human study is to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of increasing doses of PF-07265028 as monotherapy and in combination with sasanlimab; identify the maximum tolerated dose (MTD) of PF-07265028 monotherapy; evaluate the clinical activity of monotherapy and combination; and select the recommended dose of PF-07265028 monotherapy and in combination for potential further studies and development. The study contains 2 parts, Dose Escalation (Part 1) to determine the recommended dose of PF-07265028 as single agent and in combination, followed by Dose Expansion (Part 2) in selected tumor types at the recommended dose.

ELIGIBILITY:
Key Inclusion Criteria:

Across all cohorts:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
2. Adequate hematological, kidney and liver function
3. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
4. Resolved acute effects of any prior therapy
5. All participants must provide archival formalin-fixed paraffin-embedded (FFPE) tumor tissue:

Part 1: If archival sample is older than 6 months, the participant must consent to undergo a fresh biopsy during the screening.

Part 2 Fresh tumor biopsy during screening is required unless there is archival tissues less than 3 months old and subsequent to the last systemic anti-cancer therapy.

Part 1A Monotherapy:

Histologically or cytologically confirmed advanced or metastatic solid tumors which have progressed following systemic anticancer therapies, or are resistant to standard therapy or for which no standard therapy is available, or for whom standard therapy is not tolerated.

Part 1B Combination Therapy:

Histologically or cytologically confirmed advanced or metastatic solid tumor which have progressed following systemic anticancer therapies, including at least 1 checkpoint inhibitor.

Part 2 Dose Expansion:

Histologically or cytologically confirmed advanced or metastatic malignancies, including gastric/Gastroesophageal junction cancer, Head and neck squamous cell carcinoma, or urothelial cancer (non-small cell lung cancer and other solid tumors may be included) who have progressed following systemic anticancer therapies, including at least 1 checkpoint inhibitor

Key Exclusion Criteria:

1. Participants with any other active malignancy within 3 years prior to enrollment
2. Participants with active autoimmune conditions or history of autoimmune diseases that may relapse
3. History of interstitial lung disease, pneumonitis (non-infectious) or uncontrolled lung diseases
4. History of prior immune-related adverse events (irAEs) Grade ≥3
5. Central nervous system metastases
6. Significant cardiac or pulmonary conditions or events within previous 6 months
7. Active, uncontrolled bacterial, fungal, or viral infection
8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PF-07265028
9. Prior administration of HPK1 inhibitor

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose-limiting toxicities (DLTs) in Dose Escalation (Part 1) | Cycle 1 (28 days)
  DLTs will be evaluated during Cycle 1 (a cycle is 28 days) in Part 1. The number of DLTs will be used to determine the optimal dose
Number of participants with adverse events (AEs) | Baseline through up to 2 years
  AEs characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0), timing, seriousness, and relationship to study therapy.
Number of participants with clinically significant laboratory abnormalities | Baseline through up to 2 years
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.
Objective response rate (ORR) in Dose Expansion (Part 2) | Baseline through up to 2 years or until disease progression
  Tumor response based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
The pharmacokinetic profile of single and multiple doses PF-07265028 alone and in combination with sasanlimab through Cmax. | Days 1, 8, 15, 16 and 22 of Cycle 1 (each cycle is 28 days)
  Maximum observed plasma concentration of PF-07265028 (Cmax) and Maximum observed steady state plasma concentration (Cmax, ss)
The pharmacokinetic profile of single and multiple doses PF-07265028 alone and in combination with sasanlimab through Tmax. | Days 1, 8, 15, 16 and 22 of Cycle 1 (each cycle is 28 days)
  Time to maximal observed plasma concentration of PF-07265028 (Tmax) and Time to reach Maximum Observed Steady State Plasma Concentration (Tmax,ss).
The pharmacokinetic profile of single and multiple doses PF-07265028 alone and in combination with sasanlimab through AUC | Days 1, 8, 15, 16 and 22 of Cycle 1 (each cycle is 28 days)
  Area under the concentration versus time curve from time zero to the last quantifiable time point prior to the next dose (AUClast) of PF-07265028 and area under the curve within one dose interval at steady state (AUCtau,ss)
The effect of food on the pharmacokinetic profile of PF-07265028 through Cmax. | Days 1, 8, 15, 16 and 22 of Cycle 1 (each cycle is 28 days)
  Maximum observed plasma concentration of PF-07265028 (Cmax) under fasted and fed conditions in the subset of participants
The effect of food on the pharmacokinetic profile of PF-07265028 through Tmax | Days 1, 8, 15, 16 and 22 of Cycle 1 (each cycle is 28 days)
  Time to maximal observed plasma concentration of PF-07265028 (Tmax) under fasted and fed conditions in the subset of participants
The effect of food on the pharmacokinetic profile of PF-07265028 through AUC | Days 1, 8, 15, 16 and 22 of Cycle 1 (each cycle is 28 days)
  Area under the concentration versus time curve from time zero to the last quantifiable time point prior to the next dose (AUClast) of PF-07265028 under fasted and fed conditions in the subset of participants
The pharmacokinetic profile of sasanlimab when given in combination with PF-07265028 through Cmin | Day 1 of cycle 1 (each cycle is 28 days), Day 1 of cycle 2, Day 1 of cycle 3, Day 1 of cycle 5 and thereafter every 6 cycles (each cycle is 28 days)
  Minimum plasma concentration (Cmin) will be calculated through the measured pre-dose plasma concentration
The immunogenicity of sasanlimab when given in combination with PF-07265028 through ADA and NAb | Day 1 of cycle 1 (each cycle is 28 days), Day 1 of cycle 2, Day 1 of cycle 3, Day 1 of cycle 5 and thereafter every 6 cycles (each cycle is 28 days)
  Incidence and titers of anti-drug antibodies (ADA) and neutralizing antibodies (NAb) against sasanlimab
The effect of PF-07265028 alone and in combination with sasanlimab on tumor immune biomarkers modulation | Baseline through up to 2 years
  Levels of intratumor T cells and PD-L1 expression in pre- and post-treatment tumor biopsies
ORR in Dose Escalation (Part 1) | From baseline through disease progression or study completion (approximately 2 years)
  Tumor response assessment based on RECIST 1.1
Time to event endpoints (DOR) in Dose Expansion (Part 2) | From baseline through disease progression or study completion (approximately 2 years)
  Duration of response (DOR) as assessed using RECIST 1.1.
Time to event endpoints (PFS) in Dose Expansion (Part 2) | From baseline through disease progression or study completion (approximately 2 years)
  Progression free survival (PFS) as assessed using RECIST 1.1.
Time to event endpoints (OS) in Dose Expansion (Part 2) | From baseline through disease progression or study completion (approximately 2 years)
  Overall survival (OS) assessed proportion of patients alive

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (10):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona
  - D&H Cancer Research Center LLC, Margate, Florida
  - Napa Research, Margate, Florida
  - University of Iowa, Iowa City, Iowa
  - START Midwest, Grand Rapids, Michigan
  - Mary Crowley Cancer Research - Medical City Hospital, Dallas, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4731001